CLINICAL TRIAL: NCT03661957
Title: Non Grafted Maxillary Sinus Floor Elevation With Simultaneous Implant Placement Versus the Use of Short Endosseous Implants
Brief Title: Non Grafted Maxillary Sinus Floor Elevation With Implant Placement Versus the Use of Short Endosseous Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Mansour, dentist-master student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: cairo university 99
Record Dates: First submitted 2018-09-02; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Primary Stability of Implants; Marginal Bone Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non grafted maxillary sinus floor elevation with implant pacem (Active Comparator)
  Interventions: Procedure: Non grafted maxillary sinus floor elevation with simultaneous implant placement
- using short dental implants for posterior atrophic maxilla (Experimental)
  Interventions: Procedure: using short dental implants for posterior atrophic maxilla

INTERVENTIONS:
Procedure: Non grafted maxillary sinus floor elevation with simultaneous implant placement — lateral window for sinus elevation ,membrane elevation ,implant placement , membrane for window closure
  Arms: Non grafted maxillary sinus floor elevation with implant pacem
Procedure: using short dental implants for posterior atrophic maxilla — placement of short dental implant with bone height below 8mm
  Arms: using short dental implants for posterior atrophic maxilla

SUMMARY:
Assessment the need for sinus floor elevation when restoring atrophic posterior maxilla or it will be enough to use of short implant

ELIGIBILITY:
Inclusion Criteria:

* Patients with partially edentulous in the posterior area of the maxilla, with a residual ridge that allowed insertion of ≤8 mm length implants.
* Both sexes.
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Sinus pathology.
* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site
* Immunodeficiency pathology, bruxism, stress situation (socially or professionally), emotional instability, and unrealistic aesthetic demands.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
primary stability | 6 months
  measuring primary stability using osstel

SECONDARY OUTCOMES:
marginal bone loss | 6 months
  measuring marginal bone loss using cone beam ct

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher Mansour, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes